CLINICAL TRIAL: NCT04087044
Title: Computerized Rotational Head Impulse Test-Vertical (crHIT-vertical)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neurolign (Industry)
Collaborators: University of Miami (Other); University of Pittsburgh (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: crHIT-vertical
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Vestibular Function Tests
Keywords: vestibular neuritis; vestibular migraine
MeSH Terms: conditions — Vestibular Neuronitis

STUDY DESIGN:
Intervention Model Description: 66 patients (30 patients with surgically confirmed unilateral loss, 15 patients with absent ice water calorics and resulting from vestibular neuritis and 21 patients with vestibular migraine) 120 controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vestibular dysfunction (Experimental): 66 patients: 30 patients with surgically confirmed unilateral loss, 15 patients with absent ice water calorics and resulting from vestibular neuritis and 21 patients with vestibular migraine
  Interventions: Device: Computerized Rotational Head Impulse Test ( crHIT)-Vertical
- Control (Other): 120 aged matched controls
  Interventions: Device: Computerized Rotational Head Impulse Test ( crHIT)-Vertical

INTERVENTIONS:
Device: Computerized Rotational Head Impulse Test ( crHIT)-Vertical — 1. Oculo-Motility and Positional Testing,
  2. Caloric Testing
  Other Names: crHIT Vertical

SUMMARY:
The purpose of this research study is to test whether a Computerized Rotational Head Impulse Test-Vertical (crHIT-vertical) is able to reliably evaluate the vertical semicircular canals in patients with vestibular dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to tolerate the placement of a set of goggles on their face
* Controls:

  1. no history of dizziness or imbalance
  2. normal responses on rotational chair testing
* Patients: persons clinically diagnosed with vestibular disorders

Exclusion Criteria:

* Pregnancy
* Neurodegenerative diseases

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of crHIT-vertical | 9 months
  How many participants are correctly identified as either having a vestibular dysfunction or being healthy controls

SECONDARY OUTCOMES:
Subject discomfort - symptoms | 9 months
  Number of subjects indicating motion sickness symptoms during the crHIT test. If motion sickness is present subjects are asked to rate the symptoms of motion sickness and severity on scale 1 to 5, where 1 is minimum and 5 is severe.
Subject discomfort - test apparatus | 9 months
  Subjects rate the comfort of chair, head rest and goggle on scale 1 to 5, where 1 is very uncomfortable and 5 very comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Hoffer, MD, Principal Investigator — University of Miami; Joseph Joseph Furman, PhD, Principal Investigator — University of Pittsburgh; Devin McCaslin,, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No